CLINICAL TRIAL: NCT02394171
Title: Health is Power: An Ecological Theory-based Health Intervention for Women of Color
Acronym: HIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Rebecca Lee, Full Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RebeccaLee
Record Dates: First submitted 2015-03-09; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Physical Activity
Keywords: Physical Activity; Social Cohesion; Intervention Development; Ethnic Minorities; Nutrition
MeSH Terms: conditions — Motor Activity | interventions — Social Cohesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity (Experimental): Women completed a physical activity group cohesion intervention which included six content intensive intervention sessions over a 24 week period that focused on specific group dynamics team building strategies to increase physical activity. A small team structure was used for peer problem solving and support throughout the intervention. Teams were given weekly physical activity goals, with slowly increasing weekly minutes milestones to gradually meet recommended amounts of physical activity. Sessions included brief instructions, team-based activities, and discussion with the entire group lead by a trained health educator. The intervention sessions ended with the health educator leading the teams in a brisk 15-minute walk.
  Interventions: Behavioral: Group Cohesion
- Fruit and Vegetable (Active Comparator): Women completed a fruit and vegetable group cohesion intervention which involved six content intensive intervention sessions over a 24 week period that focused on specific group dynamics team building strategies to increase fruit and vegetable consumption. A small team structure was used for peer problem solving and support throughout. Teams were given weekly fruit and vegetable consumption goals at each session, with slowly increasing weekly servings milestones to gradually meet recommended amounts of fruit and vegetable consumption. Sessions included brief instructions, team-based activities, and discussion with the entire group lead by a trained health educator. The intervention sessions ended with the health educator leading the teams in a fruit and vegetable taste test.
  Interventions: Behavioral: Group Cohesion

INTERVENTIONS:
Behavioral: Group Cohesion — See description in arm/group above

SUMMARY:
Health Is Power (HIP) was a community based health intervention designed to increase physical activity among women of color. It was funded by a grant from the National Cancer Institute of the National Institutes of Health. The purposes of the study were (1) to determine whether a 6 month, group cohesion intervention is more effective for increasing physical activity compared to a 6 month, group cohesion comparison targeting improving dietary habits (2) to determine whether residence in a neighborhood supportive for physical activity helped women maintain their physical activity from 6 to , and (3) to determine whether this effect was transculturally replicable.

DETAILED DESCRIPTION:
Objective Physical inactivity and poor dietary habits plague Americans as health challenges, with women of color most vulnerable to their detrimental effects. Individually focused interventions have not demonstrated lasting success, possibly due to the lack of focus on sustainable social and physical environment factors. Health Is Power (HIP) was a transcultural, community based, randomized controlled trial that investigated the effectiveness of a group cohesion intervention to increase physical activity in African American and Hispanic or Latina women in Houston and Austin, Texas and then tested whether women living in more supportive areas maintained their physical activity over time. Intervention development was guided by group dynamics principles anchored within an ecologic model. Women participated in three health assessments and a six month face to face intervention that included evidence-based behavioral methods - integrated into strategies to promote group cohesion - framed to account for environmental factors contributing to health disparities. Women participated in team building activities, environmental mapping exercises, and supervised walks or taste tests. Neighborhood contextual and environmental measures were measured to test ecologic factors that may contribute to behavioral maintenance.

ELIGIBILITY:
Inclusion criteria:

* African American or Hispanic/ Latina
* Between the ages of 25 and 60 years old
* Able to read, speak, and write in English or Spanish
* Not pregnant or planning to become pregnant within the next 12 months
* Resident of Harris or Travis County, Texas
* Not planning on moving in the next 12 months
* Physically inactive or did not do more than 30 min of physical activity per day on 3 or more days per week
* No history of medical illness or currently taking medication (could have medical waiver from physician if did not meet this)
* Willing to be randomized to either a physical activity group or a vegetable and fruit group
* Available between 5:30 and 8:00 PM on meeting dates.

Ages: 26 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 410 (Actual)
Dates: Start 2005-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity as measured by accelerometry and the International Physical Activity Questionnaire (IPAQ) | 6 months
  women were measured at baseline and 6 month
Maintenance in Physical Activity as measured by accelerometry and the International Physical Activity Questionnaire (IPAQ) | 6 months
  women were measured at 6 months and 12 months

REFERENCES:
- [Background] Smith-Ray RL, Mama S, Reese-Smith JY, Estabrooks PA, Lee RE. Improving participation rates for women of color in health research: the role of group cohesion. Prev Sci. 2012 Feb;13(1):27-35. doi: 10.1007/s11121-011-0241-6. PMID 21826476
- [Background] Soltero EG, Hernandez DC, O'Connor DP, Lee RE. Does social support mediate the relationship among neighborhood disadvantage, incivilities, crime and physical activity? Prev Med. 2015 Mar;72:44-9. doi: 10.1016/j.ypmed.2014.12.030. Epub 2015 Jan 3. PMID 25562756
- [Background] McAlexander KM, Mama SK, Medina A, O'Connor DP, Lee RE. The concordance of directly and indirectly measured built environment attributes and physical activity adoption. Int J Behav Nutr Phys Act. 2011 Jul 7;8:72. doi: 10.1186/1479-5868-8-72. PMID 21736740
- [Background] Lee RE, O'Connor DP, Smith-Ray R, Mama SK, Medina AV, Reese-Smith JY, Banda JA, Layne CS, Brosnan M, Cubbin C, McMillan T, Estabrooks PA. Mediating effects of group cohesion on physical activity and diet in women of color: health is power. Am J Health Promot. 2012 Mar-Apr;26(4):e116-25. doi: 10.4278/ajhp.101215-QUAN-400. PMID 22375580
- [Background] McAlexander KM, Mama SK, Medina AV, O'Connor DP, Lee RE. Concordance and correlates of direct and indirect built environment measurement among minority women. Am J Health Promot. 2012 Mar-Apr;26(4):239-44. doi: 10.4278/ajhp.100715-QUAN-241. PMID 22375575
- [Background] Ledoux T, Adamus-Leach H, O'Connor DP, Mama S, Lee RE. The association of binge eating and neighbourhood fast-food restaurant availability on diet and weight status. Public Health Nutr. 2015 Feb;18(2):352-60. doi: 10.1017/S1368980013003546. Epub 2014 Jan 24. PMID 24476972
- [Background] Lee RE, Mama SK, Medina AV, Reese-Smith JY, Banda JA, Layne CS, Baxter M, O'Connor DP, McNeill L, Estabrooks PA. Multiple measures of physical activity, dietary habits and weight status in African American and Hispanic or Latina women. J Community Health. 2011 Dec;36(6):1011-23. doi: 10.1007/s10900-011-9403-5. PMID 21519867
- [Background] Ledoux TA, Mama SK, O'Connor DP, Adamus H, Fraser ML, Lee RE. Home Availability and the Impact of Weekly Stressful Events Are Associated with Fruit and Vegetable Intake among African American and Hispanic/Latina Women. J Obes. 2012;2012:737891. doi: 10.1155/2012/737891. Epub 2012 May 14. PMID 22666558
- [Background] Adamus-Leach HJ, Wilson PL, O'Connor DP, Rhode PC, Mama SK, Lee RE. Depression, stress and body fat are associated with binge eating in a community sample of African American and Hispanic women. Eat Weight Disord. 2013 Jun;18(2):221-7. doi: 10.1007/s40519-013-0021-3. Epub 2013 Apr 9. PMID 23760851
- [Background] Wilson PL, O'Connor DP, Kaplan CD, Bode S, Mama SK, Lee RE. Relationship of fruit, vegetable, and fat consumption to binge eating symptoms in African American and Hispanic or Latina women. Eat Behav. 2012 Apr;13(2):179-82. doi: 10.1016/j.eatbeh.2012.01.007. Epub 2012 Jan 24. PMID 22365808
- [Background] Lee RE, Medina AV, Mama SK, Reese-Smith JY, O'Connor DP, Brosnan M, Cubbin C, McMillan T, Estabrooks PA. Health is Power: an ecological, theory-based health intervention for women of color. Contemp Clin Trials. 2011 Nov;32(6):916-23. doi: 10.1016/j.cct.2011.07.008. Epub 2011 Jul 18. PMID 21782975
- [Background] Lopez Y 3rd, O'Connor DP, Ledoux TA, Lee RE. Analysis of body composition methods in a community sample of African American women. Women Health. 2011 Nov 30;51(8):709-23. doi: 10.1080/03630242.2011.623222. PMID 22185287
- [Background] Lee RE, Mama SK, Medina AV, Ho A, Adamus HJ. Neighborhood factors influence physical activity among African American and Hispanic or Latina women. Health Place. 2012 Jan;18(1):63-70. doi: 10.1016/j.healthplace.2011.08.013. PMID 22243907
- [Background] Mama SK, Quill BE, Fernandez-Esquer ME, Reese-Smith JY, Banda JA, Lee RE. Body image and physical activity among Latina and African American women. Ethn Dis. 2011 Summer;21(3):281-7. PMID 21942159
- [Background] Mama SK, McNeill LH, McCurdy SA, Evans AE, Diamond PM, Adamus-Leach HJ, Lee RE. Psychosocial factors and theory in physical activity studies in minorities. Am J Health Behav. 2015 Jan;39(1):68-76. doi: 10.5993/AJHB.39.1.8. PMID 25290599